CLINICAL TRIAL: NCT01167361
Title: Epidemiology Of Respiratory Virus Infections In Children
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: XPD10-082 RESVPI
Record Dates: First submitted 2010-07-20; First posted 2010-07-22 (Estimated); Last update posted 2012-10-31 (Estimated); Status verified 2011-07

CONDITIONS: Respiratory Virus Infection
Keywords: upper respiratory tract infection; lower respiratory tract infection
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Specimens collected will include nasopharyngeal washes, nasopharyngeal swabs, tracheal aspirates and bronchoalveolar lavage as ordered by the treating physician. Diagnostic studies on this specimen will be performed as ordered and the results will be available to the treating physicians after reporting. An aliquot from the leftover sample remaining after clinical diagnostic testing will be used for FilmArrayTM analysis
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Children with upper or lower respiratory infections: Respiratory Virus infections in children who are symptomatic with either an Upper Respiratory Tract Infections and/or Lower Respiratory Tract Infections is determined by using a novel highly sensitive and rapid assay for RV detection. An aliquot from the leftover sample remaining after clinical diagnostic testing will be used for FilmArrayTM analysis. Specimens collected will include nasopharyngeal washes, nasopharyngeal swabs, tracheal aspirates and bronchoalveolar lavage as ordered by the treating physician. Diagnostic studies on this specimen will be performed as ordered and the results will be available to the treating physicians after reporting.

SUMMARY:
This study aims to prospectively estimate the incidence of Respiratory virus (RV) infections in children with symptoms of an upper respiratory tract infection (URTI) or lower respiratory tract infection (LRTI) at St. Jude Children's Research Hospital (SJCRH) using the FilmArrayTM System, a novel highly sensitive and rapid assay for RV detection. An aliquot from the leftover sample remaining after clinical diagnostic testing will be used for FilmArrayTM analysis. Patients will be accrued on the study over a one year period.

DETAILED DESCRIPTION:
The Primary Objective of the study is:

* Prospectively estimate the incidence of Respiratory virus (RV) infections in children with symptoms of an upper respiratory tract infection (URTI) or lower respiratory tract infection (LRTI) at St. Jude Children's Research Hospital(SJCRH).

The Secondary Objectives of the study are:

* Study the association between RV infections and clinical variables.
* Prospectively estimate the duration of RV infections in symptomatic children at SJCRH.
* Compare the sensitivity and specificity of the current molecular method of analysis of respiratory viruses with the FilmArrayTM method.

ELIGIBILITY:
Inclusion Criteria:

* Birth to less than or equal to 18 years.
* Patients with an URTI or LRTI undergoing collection of respiratory secretions at SJCRH, by nasopharyngeal wash, nasopharyngeal swab, tracheal aspirate or bronchoalveolar lavage as ordered by the treating physician.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with an URTI or LRTI undergoing collection of respiratory secretions at St Jude by nasopharyngeal wash, nasopharyngeal swab, tracheal aspirate or bronchoalveolar lavage as ordered by the treating physician.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2010-09; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
This study measures the incidence of Respiratory virus (RV) infections in children with symptoms of an upper respiratory tract infection (URTI) or lower respiratory tract infection (LRTI) using the FilmArray System | 1 year
  This study uses FilmArrayTM System, a novel highly sensitive and rapid assay for respiratory virus infection. An aliquot from the leftover sample remaining after clinical diagnostic testing will be used for FilmArrayTM analysis

SECONDARY OUTCOMES:
Time of first detection of the virus as related to day of transplant, Time of first detection of the virus as related to day of chemotherapy and duration of viral shedding from the time of first detection will all be measured. | 1 year
  Different variables will be collected to find the association between Respiratory virus and clinical variables
This study prospectively estimates and measures the duration of Respiratory Virus infections in symptomatic children by studying the epidemiology and natural history of infections with these viruses . | 1 year
  These viruses have been known to cause interstitial lung disease, will help clarify the etiology of "idiopathic pneumonia" post chemotherapy .
This study analyses respiratory viruses using Filmarray TM method | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ashok Srinivasan, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St . Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org